CLINICAL TRIAL: NCT04128111
Title: Study on the Correlation Between TCM Syndrome, Inflammatory Phenotype and Biomarker of Bronchial Asthma: An Observational Study
Brief Title: Study on the Correlation Between TCM Syndrome, Inflammatory Phenotype and Biomarker of Bronchial Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Collaborators: Henan Provincial People's Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: TCM syndrome of Asthma
Record Dates: First submitted 2019-09-11; First posted 2019-10-16 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-10

CONDITIONS: Bronchial Asthma
Keywords: Bronchial Asthma; TCM Syndrome; Inflammation Phenotype; Biomarker
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — 1.The inflammation phenotype will be determined by measuring the different proportions of eosinophils, neutrophils and mast cells in induced sputum.2.Indicators such as 8-isoprostaglandin, nitric oxide products and leukotrienes in exhaled breath condensate, exhaled nitric oxide, urine LTE4, and serum eosinophils, eosinophilic cationic protein, periosteal protein, IL-4, IL-5, IL-8, IL-13, IL-17, TNF-α, Eotaxin-2, total IgE and specific IgE will be measured in peripheral venous serum samples will be measured.3.Urine will be taken from 2 to 3 mL in the morning and stored at - 70°C on ice. The level of LTE4 will be determined by ELISA.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute Exacerbation: Exacerbations of asthma are episodes characterized by a progressive increase in symptoms of shortness of breath, cough, wheezing or chest tightness and progressive decrease in lung function, i.e. they represent a change from the patient's usual status that is sufficient to require a change in treatment.
- Non-acute exacerbation: Non-acute exacerbation of asthma includes chronic remission and clinical delays.Clinical remission stage refers to an absence of wheezing, chest tightness, cough and other symptoms for more than 1 year.Chronic duration refers to that symptoms, such as wheezing, chest tightness, cough and so on, attack at different frequency and different degrees every week.
- Healthy Volunteer: Health is not only the absence of disease or infirmity, but also a state of physical, mental, and social perfection.

SUMMARY:
This study aims to determine the TCM syndrome pattern and the distribution of inflammation phenotype in different stages of bronchial asthma; to explore the correlation between TCM syndrome and inflammation phenotype. Secondly screening biomarkers that can be recognized by TCM syndromes and inflammatory phenotypes of bronchial asthma, and provide a basis for individualized diagnosis and treatment of diseases.

DETAILED DESCRIPTION:
The clinical heterogeneity of bronchial asthma was strong.The TCM syndrome was complicated and mostly treated on stage, type, excess and deficiency.The phenotype was numerous and more classified from inflammation type, clinical classification, internal phenotype, etc.The flammatory phenotype was the more common type.The pathological basis of asthma was closely related to the infiltration of inflammatory mediators such as Airway eosinophil cells, so it was important to find the specific biomarker. The correlation between TCM syndrome, inflammatory phenotype and its biomarker wsa not clear. So we put forward theoretical hypothesis:There was of correlation between TCM syndrome and inflammatory phenotype of asthma.The biological target was contributes to the confirmation for TCM syndrome and inflammatory phenotype.The following research was planned to be carried out: relying on the registration system of National TCM Clinical Research Base to enroll in 900 cases patients in the acute and remission period of asthma and healthy physical examination crowd, filling in the patient's general demographic data, disease status, lung function, TCM syndrome and score and collecting the sputum, exhaled gas, urine, peripheral venous serum specimens and biomarker to be tested on the same day. Based on the clinical research database, confirming syndrome and in phenotype, clarifying the correlation between syndrome and phenotype and selecting identifiable biomarker by using correlation analysis, principal component analysis, multiple regression analysis, neural network analysis and other methods.The research provided evidence for the study of the essence of syndrome and phenotype and provided evidence for individualized diagnosis and treatment of diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with definite dignosis of bronchial asthma or healthy volunteer;
2. Ages range from 18 years to 80 years old;
3. Not anticipated in other clinical studies within 1 month before enrollment;
4. Signed informed consent.

Exclusion Criteria:

1. Acute asthma exacerbation patients with respiratory failure, mechanical ventilation;
2. Patients with unconsciousness, dementia, various mental disorders;
3. Complicated with hematological malignancies , heart failure(Acute myocardial infarction, cardiac function grade 3 or above), severe liver or kidney diseases;
4. Complicated with neuromuscular disorders affecting respiratory and motor function, unable to complete the six-minute walk test;
5. People who are participating in other clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The diagnosis and staging of bronchial asthma refer to"Chinese Guideline for The Prevention and Management of Bronchial Asthma (2016 edition)"and "The Chinese experts'consensus on the evaluation and management of asthma exacerbation"by Chinese Society of Respiratory Diseases and China Asthma Alliance.
  Reference Standard for Healthy Population The Concept of "Health" by the United Nations World Health Organization (WHO).The investigators will only enroll subjects in whom above diagnosis is firmly established.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Phenotype | Each enrolled patient will be measured only once when enrollment.
  The inflammation phenotype will be determined by measuring the different proportions of eosinophils, neutrophils and mast cells in induced sputum.The inflammatory phenotypes of asthma can be divided into eosinophil asthma(eosinophil > 1.01%) ， neutrophil asthma(neutrophil > 61%)， Oligocellular asthma (eosinophil > 61%)and mixed cell asthma(eosinophil > 1.01%, neutrophil > 61%).

SECONDARY OUTCOMES:
Biomarker | Each enrolled patient will be measured only once when enrollment.
  Indicators such as 8-isoprostaglandin, nitric oxide products and leukotrienes in exhaled breath condensate, exhaled nitric oxide, urine LTE4, and serum eosinophils, eosinophilic cationic protein, periosteal protein, IL-4, IL-5, IL-8, IL-13, IL-17, TNF-α, Eotaxin-2, total IgE and specific IgE will be measured in peripheral venous serum samples will be measured.
FeNO | Each enrolled patient will be measured only once when enrollment.
  Measurement of Exhaled Nitric Oxide by Swedish NIOX.
Exhaled Breath Condensate（EBC） | Each enrolled patient will be measured only once when enrollment.
  EBC will be collected by EcoScreen, 8-isoprostaglandin, nitric oxide products and leukotrienes will be measured by ELISA.
Urine Specimen | Each enrolled patient will be measured only once when enrollment.
  Urine will be taken from 2 to 3 mL in the morning and stored at - 70°C on ice. The level of LTE4 will be determined by ELISA.
Peripheral Venous Serum Specimens | Each enrolled patient will be measured only once when enrollment.
  In the morning, 10ml of elbow vein blood will be extracted on an empty stomach, centrifuged at 3000rpm for 5min, and serum will be separated and stored at - 70 ℃. Serum eosinophils, eosinophil cationic protein, periosteal protein, total IgE , specific IgE, cytokines IL-4, IL-5, IL-8, IL-13, IL-17, TNF - α, eotaxin-2, etc. will be measured. All the procedures will be described according to the kit. Ming Shu operation.
TCM Syndrome | Each enrolled patient will be measured only once when enrollment.
  According to the comprehensive analysis of four TCM diagnostic methods, the syndrome differentiation will be determined.
General demographic data | Each enrolled patient will be measured only once when enrollment.
  General demographic data, including name, age（years）, sex(male / female), BMI(kg/m2), occupation, smoking history (years)and drinking history(years), will be recorded.
Disease Conditions | Each enrolled patient will be measured only once when enrollment.
  The course of disease, number of acute attack，having a cold, disease-related hospitalizatation past year and drug use situations including glucocorticoid and bronchial diastole.
Asthma Control Test (ACT) Scores | Each enrolled patient will be measured only once when enrollment.
  ACT includes five questions. Every question will be assessed using a 5-point scale with scores ranging from 5 to 25. The higher the score, the better the symptom control.25 is considered complete control level, 20 ~ 24 is considered good control level, and <20 is considered non-control level.
ACQ-5 Scores | Each enrolled patient will be measured only once when enrollment.
  There are seven questions, with a score of 0-6 in every question.The final ACQ score consists of the average score of the seven questions.The higher the score, the worse the symptom control. A score of 0 ~ 0.75 means ideal asthma control; 0.75 ~ 1.5 is the "gray" area;> 1.5 indicates poor control.
Lung function and diurnal variation rate of PEF | Each enrolled patient will be measured only once when enrollment.
  Forced vital capacity (FVC), forced expiratory volume in one second (FEV1), the percentage of FEV1 in the estimated value, and the diurnal variation rate of PEF will be measured.
6-minute walk test | Each enrolled patient will be measured only once when enrollment.
  6-minute walking distance will be measured.Reference to American Thoracic Society Six-minute walking test will be conducted on all subjects in the published Six-minute Walking Guidelines, and the six-minute walking distance will be measured.
Acute Exacerbations | Each enrolled patient will be measured only once when enrollment.
  The number, causes, treatment place, medications, costs and outcomes of acute exacerbations will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Suyun Li, Professor, Study Director — The First Affiliated Hospital of Henan University of Chinese Medicine
Locations (1):
- The First Affiliated Hospital of Henan University of Traditional Chinese Medicine, Zhengzhou, Henan, China